CLINICAL TRIAL: NCT00100048
Title: Multicenter, Double-Blind, Randomized, Dose Ranging Study to Compare the Safety and Activity of MK0518 Plus Tenofovir and Lamivudine (3TC) Versus Efavirenz Plus Tenofovir and Lamivudine (3TC) in ART-Naive, HIV-Infected Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of an Investigational Drug in HIV Infected Patients (0518-004)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-004; 2004_096
Record Dates: First submitted 2004-12-22; First posted 2004-12-23 (Estimated); Results first posted 2010-03-29 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 600 mg monotherapy (Experimental): MK0518 600 mg twice daily
  Interventions: Drug: Comparator: MK0518 monotherapy
- 400 mg monotherapy (Experimental): MK0518 400 mg twice daily
  Interventions: Drug: Comparator: MK0518 monotherapy
- 200 mg monotherapy (Experimental): MK0518 200 mg twice daily
  Interventions: Drug: Comparator: MK0518 monotherapy
- 100 mg monotherapy (Experimental): MK0518 100 mg twice daily
  Interventions: Drug: Comparator: MK0518 monotherapy
- placebo monotherapy (Placebo Comparator): Placebo to MK0518 twice daily
  Interventions: Drug: Placebo monotherapy
- 600 mg combo therapy (Experimental): MK0518 600 mg + tenofovir + lamivudine
  Interventions: Drug: Comparator: MK0518 combination therapy; Drug: Comparator: tenofovir; Drug: Comparator: lamivudine
- 400 mg combo therapy (Experimental): MK0518 400 mg + tenofovir + lamivudine
  Interventions: Drug: Comparator: MK0518 combination therapy; Drug: Comparator: tenofovir; Drug: Comparator: lamivudine
- 200 mg combo therapy (Experimental): MK0518 200 mg + tenofovir + lamivudine
  Interventions: Drug: Comparator: MK0518 combination therapy; Drug: Comparator: tenofovir; Drug: Comparator: lamivudine
- 100 mg combo therapy (Experimental): MK0518 100 mg + tenofovir + lamivudine
  Interventions: Drug: Comparator: MK0518 combination therapy; Drug: Comparator: tenofovir; Drug: Comparator: lamivudine
- EFV combo therapy (Active Comparator): efavirenz + tenofovir + lamivudine
  Interventions: Drug: Comparator: efavirenz; Drug: Comparator: tenofovir; Drug: Comparator: lamivudine

INTERVENTIONS:
Drug: Comparator: MK0518 monotherapy — MK0518 twice daily for 10 days
  Arms: 100 mg monotherapy; 200 mg monotherapy; 400 mg monotherapy; 600 mg monotherapy
Drug: Comparator: MK0518 combination therapy — MK0518 twice daily for 48 weeks
  Arms: 100 mg combo therapy; 200 mg combo therapy; 400 mg combo therapy; 600 mg combo therapy
Drug: Comparator: efavirenz — efavirenz 600 mg every night at bedtime for 48 weeks
  Arms: EFV combo therapy
Drug: Comparator: tenofovir — tenofovir 300 mg daily for 48 weeks
  Arms: 100 mg combo therapy; 200 mg combo therapy; 400 mg combo therapy; 600 mg combo therapy; EFV combo therapy
Drug: Comparator: lamivudine — lamivudine 300 mg daily for 48 weeks
  Arms: 100 mg combo therapy; 200 mg combo therapy; 400 mg combo therapy; 600 mg combo therapy; EFV combo therapy
Drug: Placebo monotherapy — Placebo to MK0518 twice daily
  Arms: placebo monotherapy

SUMMARY:
This is a study that will investigate the safety and efficacy of an investigational drug in Human immunodeficiency virus (HIV) infected patients.

DETAILED DESCRIPTION:
Participants who completed 48 weeks of the original 48-week double-blind study were invited to continue in two extensions: MK0518-004-10 (NCT00100048), which extended the study to 144 weeks, and MK0518-004-20 (NCT00100048), which extended the study to 240 weeks. Participants who had been randomized to MK0518 in the base study continued at 400 mg MK0518 twice daily.

Participants randomized to efavirenz in the base study continued to receive efavirenz at the dosage given in the base study. The doses of open label tenofovir and lamivudine continued unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be HIV positive who must have received less than 7 days total of any antiretroviral therapy (HIV related therapy)

Extension Studies:

* First extension: Patient completed the 48-week base study
* Second extension: Patient completed the first 144-week extension study

Exclusion Criteria:

* Less than 18 years of age
* Individuals who currently do not test positive for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2005-01; Primary Completion 2006-10 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Markowitz M, Morales-Ramirez JO, Nguyen BY, Kovacs CM, Steigbigel RT, Cooper DA, Liporace R, Schwartz R, Isaacs R, Gilde LR, Wenning L, Zhao J, Teppler H. Antiretroviral activity, pharmacokinetics, and tolerability of MK-0518, a novel inhibitor of HIV-1 integrase, dosed as monotherapy for 10 days in treatment-naive HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2006 Dec 15;43(5):509-15. doi: 10.1097/QAI.0b013e31802b4956. PMID 17133211
- [Background] Murray JM, Emery S, Kelleher AD, Law M, Chen J, Hazuda DJ, Nguyen BY, Teppler H, Cooper DA. Antiretroviral therapy with the integrase inhibitor raltegravir alters decay kinetics of HIV, significantly reducing the second phase. AIDS. 2007 Nov 12;21(17):2315-21. doi: 10.1097/QAD.0b013e3282f12377. PMID 18090280
- [Background] Markowitz M, Nguyen BY, Gotuzzo E, Mendo F, Ratanasuwan W, Kovacs C, Prada G, Morales-Ramirez JO, Crumpacker CS, Isaacs RD, Gilde LR, Wan H, Miller MD, Wenning LA, Teppler H; Protocol 004 Part II Study Team. Rapid and durable antiretroviral effect of the HIV-1 Integrase inhibitor raltegravir as part of combination therapy in treatment-naive patients with HIV-1 infection: results of a 48-week controlled study. J Acquir Immune Defic Syndr. 2007 Oct 1;46(2):125-33. doi: 10.1097/QAI.0b013e318157131c. PMID 17721395
- [Background] Markowitz M, Nguyen BY, Gotuzzo E, Mendo F, Ratanasuwan W, Kovacs C, Prada G, Morales-Ramirez JO, Crumpacker CS, Isaacs RD, Campbell H, Strohmaier KM, Wan H, Danovich RM, Teppler H; Protocol 004 Part II Study Team. Sustained antiretroviral effect of raltegravir after 96 weeks of combination therapy in treatment-naive patients with HIV-1 infection. J Acquir Immune Defic Syndr. 2009 Nov 1;52(3):350-6. doi: 10.1097/QAI.0b013e3181b064b0. PMID 19648823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary therapy period:
  For Part I (10 day monotherapy): 24-Jan-2005 to 04-May-2005
  Part II (Dose Ranging): 14-Jun-2005 to 04-Oct-2006 (48 weeks); 14-Jun-2005 to 12-Jul-2010 (240 weeks)
  Multicenter (29) in the United States (14) and Ex-US (15)
Pre-assignment Details: Patients with Human Immunodeficiency Virus (HIV) Ribonucleic acid (RNA) of at least 5000 copies/mL and cluster of differentiation 4 (CD4) cell counts of at least 100 cells/mm3. All patients must have met laboratory criteria.
  206 enrolled; 5 from Cohort I did not continue to the combination phase. Therefore 201 entered the combination phase.
Groups:
- MK0518 100 mg b.i.d.: Cohort I-Monotherapy Phase
  MK0518 100 mg twice daily (b.i.d.)
  Cohort II Combined-Combination Therapy Phase
  MK0518 100 mg + tenofovir + lamivudine
- MK0518 200 mg b.i.d: Cohort I-Monotherapy Phase
  MK0518 200 mg b.i.d
  Cohort II Combined-Combination Therapy Phase
  MK0518 200 mg + tenofovir + lamivudine
- MK0518 400 mg b.i.d.: Cohort I-Monotherapy Phase
  MK0518 400 mg b.i.d.
  Cohort II Combined-Combination Therapy Phase
  MK0518 400 mg + tenofovir + lamivudine
- MK0518 600 mg b.i.d.: Cohort I-Monotherapy Phase
  MK0518 600 mg b.i.d.
  Cohort II Combined-Combination Therapy Phase
  MK0518 600 mg + tenofovir + lamivudine
- Placebo: Cohort I-Monotherapy Phase
  Placebo to MK0518 b.i.d.
- Efavirenz 600 mg q.h.s.: Cohort II Combined-Combination Therapy Phase
  efavirenz 600 mg every night at bedtime (q.h.s.)
Period: Cohort I-Monotherapy Phase 10 Days
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo | Efavirenz 600 mg q.h.s.
Started | 7 | 7 | 6 | 8 | 7 | 0 (participants only assigned Efavirenz 600 mg q.h.s in Cohort II Combined-Combination Therapy Phase)
Treated | 7 | 7 | 6 | 8 | 7 | 0
Completed | 7 (7 Subjects Continued to Cohort II Combined-Combination Therapy Phase (48 Weeks)) | 7 (7 Subjects Continued to Cohort II Combined-Combination Therapy Phase (48 Weeks)) | 6 (6 Subjects Continued to Cohort II Combined-Combination Therapy Phase (48 Weeks)) | 8 (6 Subjects Continued to Cohort II Combined-Combination Therapy Phase (48 Weeks)) | 7 (4 Subjects Continued to Cohort II, as part of the Efavirenz 600 mg q.d. arm) | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort I & II-Combination Therapy Phase
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo | Efavirenz 600 mg q.h.s.
Started | 41 (7 subjects from the Monotherapy Phase and 34 new subjects) | 40 (7 subjects from the Monotherapy Phase and 33 new subjects) | 41 (6 subjects from the Monotherapy Phase and 35 new subjects) | 40 (8 subjects from the Monotherapy Phase and 32 new subjects) | 0 (participants only assigned Placebo in Cohort I-Monotherapy Phase.) | 39 (4 subjects from the Monotherapy Phase (Placebo)and 35 new subjects)
Treated | 39 | 40 | 41 | 40 | 0 | 38
Never Treated | 2 (Randomised in Cohort II did not start Period) | 0 | 0 | 0 | 0 | 1 (Randomised in Cohort II did not start Period)
Completed | 27 | 31 | 28 | 30 | 0 | 26
Not Completed | 14 | 9 | 13 | 10 | 0 | 13
Not completed — Never Treated | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 3 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 3 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 5 | 0 | 4
Not completed — Other Reason | 7 | 1 | 4 | 2 | 0 | 0
Not completed — Completed Base Study, Did Not Continue | 1 | 1 | 2 | 0 | 0 | 2
Not completed — Laboratory Adverse Experience | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK0518 100 mg b.i.d.: Cohort I-Monotherapy Phase (10 Days)
  MK0518 100 mg twice daily (b.i.d.)
  Cohort II Combined-Combination Therapy Phase (48 Weeks) MK0518 100 mg b.i.d
- MK0518 200 mg b.i.d: Cohort I-Monotherapy Phase (10 Days)
  MK0518 200 mg b.i.d
  Cohort II Combined-Combination Therapy Phase (48 Weeks) MK0518 200 mg + tenofovir + lamivudine
- MK0518 400 mg b.i.d.: Cohort I-Monotherapy Phase (10 Days)
  MK0518 400 mg b.i.d.
  Cohort II Combined-Combination Therapy Phase (48 Weeks) MK0518 400 mg + tenofovir + lamivudine
- MK0518 600 mg b.i.d.: Cohort I-Monotherapy Phase (10 Days)
  MK0518 600 mg b.i.d.
  Cohort II Combined-Combination Therapy Phase (48 Weeks) MK0518 600 mg + tenofovir + lamivudine
- Placebo / Efavirenz 600 mg Once Daily (q.d.): Cohort I-Monotherapy Phase (10 Days)
  Placebo to MK0518 b.i.d.
  Cohort II Combined-Combination Therapy Phase (48 Weeks)
  Efavirenz + Tenofovir + Lamivudine
- Total: Total of all reporting groups
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo / Efavirenz 600 mg Once Daily (q.d.) | Total
Number analyzed (Participants) | 41 | 40 | 41 | 42 | 42 | 206
Age, Continuous [Mean (Full Range); unit: Years] — Cohort I Participants: MK0518 100 mg b.i.d. (7); MK0518 200 mg b.i.d. (7); MK0518 400 mg b.i.d. (6); MK0518 600 mg b.i.d. (8); Placebo Cohort (7)
  Cohort II Participants: MK0518 100 mg b.i.d. (33); MK0518 200 mg b.i.d. (33); MK0518 400 mg b.i.d. (35); MK0518 600 mg b.i.d. (34); Efavirenz 600 mg q.d. (34)
  Cohort I & II Participants Combined: MK0518 100 mg b.i.d. (39); MK0518 200 mg b.i.d. (40); MK0518 400 mg b.i.d. (41); MK0518 600 mg b.i.d. (40); Efavirenz 600 mg q.d. (38)
  Years
    Cohort I | 46 [31 to 68] | 37 [22 to 57] | 41 [25 to 55] | 39 [30 to 49] | 36 [21 to 51] | 40 [21 to 68]
    Cohort II | 34 [19 to 58] | 31 [21 to 56] | 34 [19 to 50] | 36 [20 to 49] | 36 [22 to 54] | 35 [19 to 58]
    Cohort I & II Combined | 37 [19 to 68] | 34 [21 to 57] | 36 [19 to 55] | 37 [20 to 49] | 36 [22 to 54] | 36 [19 to 68]
Sex/Gender, Customized [Number; unit: participants]
  Female (Cohort I) | 0 | 1 | 0 | 0 | 1 | 2
  Male (Cohort I) | 7 | 6 | 6 | 8 | 6 | 33
  Female (Cohort II) | 6 | 10 | 4 | 11 | 8 | 39
  Male (Cohort II) | 27 | 23 | 31 | 23 | 26 | 130
  Never Treated Cohort II | 1 | 0 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White (Cohort I) | 4 | 4 | 3 | 8 | 3 | 22
  Black (Cohort I) | 1 | 1 | 0 | 0 | 0 | 2
  Asian (Cohort I) | 0 | 0 | 0 | 0 | 1 | 1
  Hispanic (Cohort I) | 2 | 2 | 3 | 0 | 3 | 10
  White (Cohort II) | 4 | 10 | 11 | 8 | 10 | 43
  Black (Cohort II) | 1 | 1 | 1 | 0 | 0 | 3
  Asian (Cohort II) | 3 | 6 | 8 | 7 | 8 | 32
  Hispanic (Cohort II) | 12 | 9 | 10 | 9 | 10 | 50
  Other (Cohort II) | 13 | 7 | 5 | 10 | 6 | 41
  Never Treated (Cohort II) | 1 | 0 | 0 | 0 | 1 | 2
Cluster of differentiation 4 (CD4) Cell Count [Mean (Full Range); unit: cells/mm^3] — Cohort I Participants: MK0518 100 mg b.i.d. (7); MK0518 200 mg b.i.d. (7); MK0518 400 mg b.i.d. (6); MK0518 600 mg b.i.d. (8); Placebo Cohort (7) Cohort II Participants: MK0518 100 mg b.i.d. (33); MK0518 200 mg b.i.d. (33); MK0518 400 mg b.i.d. (35); MK0518 600 mg b.i.d. (34); Efavirenz 600 mg q.d. (34) Cohort I & II Participants Combined: MK0518 100 mg b.i.d. (39); MK0518 200 mg b.i.d. (40); MK0518 400 mg b.i.d. (41); MK0518 600 mg b.i.d. (40); Efavirenz 600 mg q.d. (38)
  cells/mm^3
    Cohort I | 415 [138 to 745] | 343 [149 to 624] | 256 [96 to 602] | 569 [241 to 1034] | 343 [115 to 599] | 394 [96 to 1034]
    Cohort II | 293 [76 to 736] | 292 [70 to 723] | 348 [95 to 1017] | 245 [99 to 734] | 276 [77 to 744] | 291 [70 to 1017]
    Cohort I and II Combined | 272 [76 to 758] | 277 [70 to 723] | 293 [95 to 1017] | 244 [99 to 786] | 225 [77 to 744] | 266 [70 to 1017]
Plasma Human Immunodeficiency Virus (HIV) Ribonucleic acid (RNA) [Geometric Mean (Full Range); unit: copies/mL] — Cohort I Participants: MK0518 100 mg b.i.d. (7); MK0518 200 mg b.i.d. (7); MK0518 400 mg b.i.d. (6); MK0518 600 mg b.i.d. (8); Placebo Cohort (7) Cohort II Participants: MK0518 100 mg b.i.d. (33); MK0518 200 mg b.i.d. (33); MK0518 400 mg b.i.d. (35); MK0518 600 mg b.i.d. (34); Efavirenz 600 mg q.d. (34) Cohort I & II Participants Combined: MK0518 100 mg b.i.d. (39); MK0518 200 mg b.i.d. (40); MK0518 400 mg b.i.d. (41); MK0518 600 mg b.i.d. (40); Efavirenz 600 mg q.d. (38)
  copies/mL
    Cohort I | 44989 [3890 to 225000] | 34143 [5420 to 168000] | 37728 [6850 to 152000] | 93911 [17100 to 388000] | 58412 [7630 to 456000] | 51496 [3890 to 456000]
    Cohort II | 65982 [4200 to 750000] | 73646 [7490 to 750000] | 47019 [2440 to 499000] | 61929 [3450 to 750000] | 76752 [7500 to 675000] | 63965 [2440 to 750000]
    Cohort I and II Combined | 58206 [4200 to 750000] | 64715 [7490 to 750000] | 43083 [2440 to 499000] | 57919 [3450 to 750000] | 67554 [3340 to 675000] | 57437 [2440 to 750000]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) on Day 10 (Cohort I)
Description: Mean change from baseline on Day 10 in plasma Human Immunodeficiency Virus (HIV) Ribonucleic acid (RNA) (copies/mL)
Time Frame: Baseline and Day 10
Population: The analysis population is based upon the modified intent to treat (MITT) approach, where patients are included in the treatment group to which they were randomized. Patients who were randomized but never dosed are not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: copies/mL
Groups:
- MK0518 100 mg b.i.d.: Cohort I-Monotherapy Phase
  MK0518 100 mg twice daily (b.i.d.)
- MK0518 200 mg b.i.d: Cohort I-Monotherapy Phase
  MK0518 200 mg b.i.d
- MK0518 400 mg b.i.d.: Cohort I-Monotherapy Phase
  MK0518 400 mg b.i.d.
- MK0518 600 mg b.i.d.: Cohort I-Monotherapy Phase
  MK0518 600 mg b.i.d.
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 7 | 7 | 6 | 8 | 7
copies/mL | -1.93 [-2.44 to -1.42] | -1.98 [-2.49 to -1.47] | -1.66 [-1.99 to -1.34] | -2.16 [-2.55 to -1.77] | -0.17 [-0.42 to 0.07]

2. Primary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs) and Number of Patients With Serious CAEs at Day 10 (Cohort I)
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product.
  Serious CAEs are any AEs occurring at any dose that; Results
  in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or
  prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an
  overdose.
Time Frame: 10 days
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | Placebo
Number analyzed (Participants) | 7 | 7 | 6 | 8 | 7
participants
  With CAEs | 4 | 2 | 3 | 5 | 5
  Without CAEs | 3 | 5 | 3 | 3 | 2
  With Serious CAEs | 0 | 0 | 0 | 0 | 0
  Without Serious CAEs | 7 | 7 | 6 | 8 | 7

3. Primary Outcome: Number of Participants With HIV RNA Levels Below 400 Copies/mL at Week 24 (Cohort II)
Time Frame: Week 24
Population: The analysis population is based upon the modified intent to treat (MITT) approach, where patients are included in the treatment group to which they were randomized. Patients who were randomized but never dosed are not included in the analysis.
  All patients who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: participants
Groups:
- MK0518 100 mg b.i.d.: Cohort II Combined-Combination Therapy Phase
  MK0518 100 mg + tenofovir + lamivudine
- MK0518 200 mg b.i.d: Cohort II Combined-Combination Therapy Phase
  MK0518 200 mg + tenofovir + lamivudine
- MK0518 400 mg b.i.d.: Cohort II Combined-Combination Therapy Phase
  MK0518 400 mg + tenofovir + lamivudine
- MK0518 600 mg b.i.d.: Cohort II Combined-Combination Therapy Phase
  MK0518 600 mg + tenofovir + lamivudine
- EFV Combo Therapy: EFV Combo Therapy Phase - Cohort II efavirenz + tenofovir +
  lamivudine
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 33 | 33 | 35 | 34 | 34
participants | 31 | 27 | 35 | 32 | 32

4. Primary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs)
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product.
Time Frame: 48 weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Groups:
- EFV Combo Therapy: EFV Combo Therapy Phase - Cohort II
  efavirenz 600 mg daily at bedtime (qhs) + tenofovir + lamivudine
  This arm included participants from Cohort I who were randomized to placebo.
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With CAEs | 31 | 35 | 36 | 35 | 34
  Without CAEs | 8 | 5 | 5 | 5 | 4

5. Other Pre Specified Outcome: Number of Participants With HIV RNA Levels Below 400 Copies/mL at Week 48
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants | 38 | 34 | 40 | 36 | 33

6. Other Pre Specified Outcome: Number of Patients With Drug-related CAEs
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs
Time Frame: 48 weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With drug-related CAEs | 18 | 20 | 19 | 19 | 27
  Without drug-related CAEs | 21 | 20 | 22 | 21 | 11

7. Other Pre Specified Outcome: Number of Patients With Serious Drug-related CAEs
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose. Drug-related are as assessed by an investigator who is a qualified physician according to his/her best clinical judgment.
Time Frame: 48 Weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With Serious drug-related CAEs | 0 | 0 | 0 | 0 | 0
  Without Serious drug-related CAEs | 39 | 40 | 41 | 40 | 38

8. Other Pre Specified Outcome: Number of Patients That Discontinued With CAEs
Time Frame: 48 Weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  Discontinued with CAEs | 0 | 0 | 0 | 0 | 0
  Did Not Discontinue with CAEs | 39 | 40 | 41 | 40 | 38

9. Other Pre Specified Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs)
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 48 Weeks
Population: The analysis population is based upon the All
  Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With LAEs | 8 | 7 | 11 | 5 | 8
  Without LAEs | 31 | 33 | 30 | 35 | 30

10. Other Pre Specified Outcome: Number of Patients With Serious LAEs
Description: Serious LAEs are any LAEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 48 Weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With serious LAEs | 0 | 0 | 0 | 0 | 0
  Without serious LAEs | 39 | 40 | 41 | 40 | 38

11. Other Pre Specified Outcome: Number of Patients With Drug-related LAEs
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) LAEs
Time Frame: 48 Weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With drug-related LAEs | 3 | 6 | 4 | 2 | 3
  Without drug-related LAEs | 36 | 34 | 37 | 38 | 35

12. Other Pre Specified Outcome: Number of Patients With Serious Drug-related LAEs
Description: as for outcome 10
Time Frame: 48 Weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With serious LAEs | 0 | 0 | 0 | 0 | 0
  Without serious LAEs | 39 | 40 | 41 | 40 | 38

13. Primary Outcome: Number of Patients With Serious CAEs (Cohort I and II Combined)
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 48 weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d. | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  With Serious CAEs | 2 | 5 | 0 | 2 | 2
  Without Serious CAEs | 37 | 35 | 41 | 38 | 36

14. Primary Outcome: Number of Patients With Serious CAEs and Non-serious CAEs at Week 144
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
  An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 144 Weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Groups:
- MK0518 b.i.d.: Cohort I-Monotherapy Phase (10 Days) MK0518 100, 200, 400, or 600 mg b.i.d.
  Cohort II Combined-Combination Therapy Phase MK0518 100, 200, 400, or 600 mg + tenofovir + lamivudine
Arm/Group | MK0518 b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 160 | 38
participants
  With CAEs | 153 | 35
  Without CAEs | 7 | 3
  With serious CAEs | 18 | 4
  Without serious CAEs | 142 | 34

15. Secondary Outcome: Number of Participants With HIV RNA Levels Below 50 Copies/mL at Week 24 (Cohort II)
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 33 | 33 | 35 | 34 | 34
participants | 28 | 27 | 33 | 32 | 31

16. Primary Outcome: Number of Participants With Clinical Adverse Experiences (AEs)and Serious Adverse Experiences (SAEs)
Description: An AE was defined as any unfavorable & unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to its use. Any worsening of a preexisting condition which was temporally associated with the use of the study drug, was also an AE.
  A SAE was any AE that resulted in death, was life threatening, resulted in a persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was cancer, or was an overdose.
Time Frame: Week 240
Population: The analysis population was based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: Participants
Groups:
- MK-0518 b.i.d.: Cohort I-Monotherapy Phase (10 Days) MK0518 100, 200, 400, or 600 mg b.i.d.
  Cohort II Combined-Combination Therapy Phase (48 Weeks) MK0518 100, 200, 400, or 600 mg + tenofovir + lamivudine
- EVF Combo Therapy: EFV Combo Therapy Phase - Cohort II
  efavirenz 600 mg daily at bedtime (qhs) + tenofovir + lamivudine
  This arm included participants from Cohort I who were randomized to placebo.
Arm/Group | MK-0518 b.i.d. | EVF Combo Therapy
Number analyzed (Participants) | 160 | 38
Participants
  Adverse experiences | 154 | 35
  Serious adverse experiences | 25 | 4

17. Primary Outcome: Number of Participants With HIV RNA (Human Immunodeficiency Virus Ribonucleic Acid) Levels Below 50 Copies/mL at Week 240
Description: HIV RNA levels were determined by AMPLICOR HIV-1 Monitor™ UltraSensitive Assay.
Time Frame: Week 240
Population: Modified-Intention-to-Treat (MITT): participants were included in the treatment group to which they were randomized, regardless of adherence to the entry criteria, treatment actually received, and deviation from the protocol. Participants who were randomized but never dosed were not included in the analyses.
Measure: Number; unit: Participants
Arm/Group | MK-0518 b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 160 | 38
Participants | 110 | 24

18. Secondary Outcome: Change From Baseline in Plasma HIV RNA at Week 24 (Cohort II)
Description: Mean change from baseline at Week 24 in plasma HIV RNA (copies/mL)
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: copies/mL
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 33 | 31 | 35 | 32 | 34
copies/mL | -2.39 [-2.58 to -2.21] | -2.20 [-2.55 to -1.86] | -2.33 [-2.51 to -2.14] | -2.49 [-2.72 to -2.26] | -2.44 [-2.69 to -2.19]

19. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Count at Week 24 (Cohort II)
Description: Mean change from baseline at Week 24 in CD4 Cell Count (cells/mm3)
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cells/mm3
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 33 | 31 | 34 | 31 | 32
cells/mm3 | 184 [144.4 to 223.6] | 122 [73.7 to 169.2] | 147 [112.3 to 182.6] | 134 [100.8 to 166.3] | 101 [59.6 to 142.8]

20. Secondary Outcome: Number of Patients With HIV RNA Level Below 50 Copies/mL and HIV RNA Level Below 400 Copies/mL at Week 96
Time Frame: 96 Weeks
Population: The analysis population is based upon the modified intent to treat (MITT) approach, where patients are included in the treatment group to which they were randomized. Patients who were randomized but never dosed are not included in the analysis. All patients switched to MK0518 400 mg b.i.d post 48 weeks.
Measure: Number; unit: participants
Arm/Group | MK0518 b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 160 | 38
participants
  HIV RNA <50 copies/mL | 133 | 32
  HIV RNA <400 copies/mL | 135 | 32

21. Secondary Outcome: Change From Baseline in Plasma HIV RNA at Week 96
Time Frame: Baseline and Week 96
Population: as for outcome 20
Measure: Mean (95% Confidence Interval); unit: copies/mL
Arm/Group | MK0518 b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 144 | 35
copies/mL | -2.30 [-2.42 to -2.19] | -2.28 [-2.57 to -2.00]

22. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline and Week 96
Population: as for outcome 20
Measure: Mean (95% Confidence Interval); unit: cells/mm3
Arm/Group | MK0518 b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 143 | 35
cells/mm3 | 221.2 [196.8 to 245.7] | 232.4 [179.6 to 285.2]

23. Secondary Outcome: Number of Participants With HIV RNA Levels Below 400 Copies/mL at Week 240
Description: HIV RNA levels were determined by AMPLICOR HIV-1 Monitor™ Standard Assay.
Time Frame: Week 240
Population: as for outcome 17
Measure: Number; unit: Participants
Arm/Group | MK-0518 b.i.d. | EVF Combo Therapy
Number analyzed (Participants) | 160 | 38
Participants | 115 | 25

24. Secondary Outcome: Change From Baseline in Plasma HIV RNA at Week 240
Description: HIV RNA levels were determined by AMPLICOR HIV-1 Monitor™ Standard Assay.
Time Frame: Baseline and Week 240
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: Log10Copies/mL
Arm/Group | MK-0518 b.i.d. | EVF Combo Therapy
Number analyzed (Participants) | 123 | 31
Log10Copies/mL | -2.29 [-2.43 to -2.15] | -2.07 [-2.45 to -1.69]

25. Secondary Outcome: Change From Baseline in CD4 (T-helper) Cell Count at Week 240
Description: Change in number of CD4 cells/mm^3 from baseline to Week 240.
Time Frame: Baseline and Week 240
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | MK-0518 b.i.d. | EVF Combo Therapy
Number analyzed (Participants) | 123 | 31
cells/mm^3 | 301.7 [268.0 to 335.5] | 275.6 [209.9 to 341.3]

26. Other Pre Specified Outcome: Number of Patients That Discontinued With LAEs
Time Frame: 48 Weeks
Population: The analysis population is based upon the All Patients As Treated (APaT) approach.
Measure: Number; unit: participants
Arm/Group | MK0518 100 mg b.i.d. | MK0518 200 mg b.i.d | MK0518 400 mg b.i.d. | MK0518 600 mg b.i.d. | EFV Combo Therapy
Number analyzed (Participants) | 39 | 40 | 41 | 40 | 38
participants
  Discontinued With LAEs | 0 | 0 | 0 | 1 | 0
  Did Not Discontinue With LAEs | 39 | 40 | 41 | 39 | 38

ADVERSE EVENTS:
Groups:
- MK-0518 b.i.d.: Cohort I-Monotherapy Phase (10 Days) MK0518 100, 200, 400, or 600 mg b.i.d.
  Cohort II Combined-Combination Therapy Phase MK0518 100, 200, 400, or 600 mg + tenofovir + lamivudine
- Efavirenz: EFV Combo Therapy Phase - Cohort II
  efavirenz 600 mg daily at bedtime (qhs) + tenofovir + lamivudine
  This arm included participants from Cohort I who were randomized to placebo.
Arm/Group | MK-0518 b.i.d. | Efavirenz
Serious Adverse Events (participants affected / at risk) | 25/160 | 4/38
Other Adverse Events (participants affected / at risk) | 147/160 | 35/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0518 b.i.d. (N=160) | Efavirenz (N=38)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kaposi's sarcoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (2) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0518 b.i.d. (N=160) | Efavirenz (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Conjunctivitis (Eye disorders) | 7 (8) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 42 (67) | 10 (19)
Flatulence (Gastrointestinal disorders) | 11 (12) | 1 (1)
Gastritis (Gastrointestinal disorders) | 7 (8) | 4 (4)
Nausea (Gastrointestinal disorders) | 35 (40) | 7 (8)
Toothache (Gastrointestinal disorders) | 9 (10) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (20) | 7 (9)
Fatigue (General disorders) | 13 (17) | 3 (4)
Influenza like illness (General disorders) | 11 (14) | 3 (3)
Malaise (General disorders) | 5 (10) | 3 (6)
Oedema peripheral (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 12 (16) | 2 (2)
Anogenital warts (Infections and infestations) | 4 (4) | 3 (4)
Body tinea (Infections and infestations) | 6 (7) | 3 (5)
Bronchitis (Infections and infestations) | 23 (31) | 2 (3)
Gastroenteritis (Infections and infestations) | 7 (10) | 2 (7)
Herpes simplex (Infections and infestations) | 10 (12) | 0 (0)
Herpes zoster (Infections and infestations) | 9 (9) | 6 (6)
Influenza (Infections and infestations) | 3 (3) | 4 (6)
Localised infection (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 30 (57) | 8 (13)
Onychomycosis (Infections and infestations) | 5 (7) | 4 (5)
Pharyngitis (Infections and infestations) | 19 (21) | 2 (3)
Sinusitis (Infections and infestations) | 16 (19) | 2 (5)
Syphilis (Infections and infestations) | 9 (10) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 39 (74) | 10 (13)
Joint sprain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 13 (29) | 4 (10)
Aspartate aminotransferase increased (Investigations) | 14 (19) | 6 (7)
Blood creatine phosphokinase increased (Investigations) | 8 (12) | 4 (5)
Blood triglycerides increased (Investigations) | 4 (8) | 2 (5)
Weight decreased (Investigations) | 3 (3) | 2 (2)
Overweight (Metabolism and nutrition disorders) | 9 (10) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (17) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (23) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 3 (4)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 2 (3)
Disturbance in attention (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 29 (33) | 13 (15)
Headache (Nervous system disorders) | 33 (56) | 16 (31)
Lethargy (Nervous system disorders) | 3 (3) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 13 (13) | 8 (9)
Anxiety (Psychiatric disorders) | 10 (11) | 4 (4)
Depression (Psychiatric disorders) | 20 (23) | 5 (6)
Insomnia (Psychiatric disorders) | 25 (29) | 5 (5)
Nightmare (Psychiatric disorders) | 1 (1) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (14) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 11 (14) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 8 (11) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.